CLINICAL TRIAL: NCT02307162
Title: A Phase I, Randomised, Double Blind, Placebo Controlled, 3-part Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Inhaled Doses of RPL554 Administered by Nebuliser to Healthy Male Subjects and Stable COPD Subjects.
Brief Title: SAD/MAD Study of a New Formulation of Nebulised RPL554 in Healthy Subjects and COPD Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-007-2014
Record Dates: First submitted 2014-11-30; First posted 2014-12-04 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Inflammatory Disorder of the Respiratory Tract; Chronic Obstructive Pulmonary Disorder
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dummy solution (Placebo Comparator): Nebulised suspension to be administered as either a single dose (Part A) or 11 doses over 6 days (Parts B anc C)
  Interventions: Drug: Placebo
- RPL554 suspension (Experimental): Nebulised suspension to be administered as either a single dose (Part A) or 11 doses over 6 days (Parts B anc C).
  Starting dose in Part A to be 1.5mg/mL with planned up to 2 fold increments. Doses in Part B will be selected from Part A. Doses in Part C to be selected from Part B
  Interventions: Drug: RPL554

INTERVENTIONS:
Drug: RPL554 — Phosphodiesterase 3 and 4 Inhibitor
  Arms: RPL554 suspension
Drug: Placebo — Dummy solution
  Arms: Dummy solution

SUMMARY:
The purpose of the study is to assess the safety of single doses and multiple doses of a new formulation of RPL554 in healthy subjects and subjects with chronic obstructive pulmonary disorder.

DETAILED DESCRIPTION:
This is a randomised, double blind, placebo controlled study of a new suspension formulation of RPL554 comprising a Single Ascending Dose (SAD) phase (Part A) in healthy subjects, a Multiple Ascending Dose (MAD) phase (Part B) in healthy subjects and a MAD phase (Part C) in stable chronic obstructive pulmonary disease (COPD) subjects. Each cohort should comprise 10 subjects in a 7 active: 3 placebo ratio

Subjects will be screened in the 14 days before the first dose of study drug and have an end of study visit 4 to 10 days after the last dose of study drug.

Part A. Single Ascending Dose Study in Healthy Male Subjects aged 18-50. Each subject will receive a single dose of study drug. The starting dose will be 1.5 mg with planned escalation as 2 fold multiples unless the safety data indicates the escalation should be at smaller intervals. If RPL554 is not well tolerated at a particular dose level, the dose may be reduced for the next cohort.The decision on whether or not to escalate to each new dose level, and the dose, will be based on a formal review by the Dose Review Group (DRG).

Part B. Multiple Ascending Dose Study in Healthy Male Subjects aged 18-50. The starting dose for Part B will be determined from the data in Part A of the study. Each subject will receive the following doses of study drug and will be confined to the study centre during dosing: three doses at intervals of 8 hours on Days 1 to 5, followed by a single morning dose on Day 6.

The DRG may determine on the basis of safety or PK data that the dosing interval for subsequent cohorts will be every 12 hours, rather than every 8 hours.

Part C. Multiple Ascending Dose in moderate, stable COPD Subjects aged 40-75 Subjects will have no known significant concurrent diseases, will not have had a recent exacerbation, and will be expected to be able to withhold regular bronchodilator therapy for the duration of the treatment phase of the study. Rescue medication with ipratropium will be allowed (and its use recorded) and subjects may continue inhaled corticosteroids at a stable dose.

The dosing schedule will be the same as for Part B

Dose Escalation Procedures The decision on whether or not to escalate to each new dose level and from one part of the study to the next and the selected dose will be based on a formal review by the DRG of safety data.

The DRG will include the Principal Investigator and Sponsor's Medical Expert (and/or delegates) and will meet by teleconference to review safety data for each cohort. The DRG will review all available safety data (including adverse events [AEs], safety laboratory tests, spirometry and ECG data) collected up to 24 hours post dose for Part A, and for up to 24 hours post final dose for Parts B and C.

Data collected during the study will be entered on case report forms and transferred to a database using double entry. Blinding will be maintained until all queries are resolved and the database is locked. AEs will be summarised by study treatment and further by intensity and relationship to study treatment. The study will primarily be evaluated using descriptive statistics.

The sample size selected is not based on any formal power calculation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Males following contraception requirements, and agree not to donate sperm during study
* 12-lead ECG within normal range and no clinically significant abnormality
* Screening Holter report (minimum 18 hours) recording that is able to be evaluated for rhythm analysis which shows no abnormality which indicates a significant impairment of subject safety or which may significantly impair interpretation
* Capable of complying with all study restrictions and procedures including ability to use the study nebuliser correctly.
* Body weight ≥50 kg.
* Negative for HIV, HBV and HCV
* Negative cotinine tests prior to randomisation.

Additional Inclusion Criteria - Healthy Subjects (Parts A and B) only:

* Males aged 18 and 50 years
* Considered to be healthy
* Vital sign assessments within ranges:

  * Systolic blood pressure 90 to 140 mmHg
  * Diastolic blood pressure 50 to 90 mmHg
  * Heart rate 45 to 90 bpm
* BMI 18 and 33 kg/m2 .
* Spirometry readings (FEV1 and FVC) ≥80% of predicted normal.
* Never smoked or is ex-smoker for ≥12 months with a smoking history of <5 pack years

Additional Inclusion Criteria - COPD Subjects (Part C) only:

* Male and females aged 40 to 75 years
* If female must be of non-childbearing potential (postmenopausal or permanently sterilised)
* BMI 18 and 33 kg/m2 (inclusive).
* COPD diagnosis (defined by ATS/ERS guidelines Celli and MacNee, 2004) with symptoms compatible with COPD for at least 1 year
* As defined in GOLD guidelines 2014: Post-bronchodilator spirometry at screening:

  * Post-salbutamol FEV1/FVC ratio 0.70
  * Post-salbutamol FEV1 ≥50 % and ≤80% of predicted normal
* No current conditions that may significantly impair subject compliance, safety or influence study results.
* Vital sign assessments within ranges:

  * Systolic blood pressure 100 to 160 mmHg
  * Diastolic blood pressure 50 to 90 mmHg
  * Heart rate 45 to 90 bpm
* Clinically stable COPD in the last 4 weeks
* Chest X-ray (post anterior) at screening, or within 6 months prior to screening showing no abnormalities, which are both clinically significant and unrelated to COPD.
* Meet the concomitant medication restrictions
* An ex-smoker for ≥6 months with a smoking history of ≥10 pack years
* Capable of withdrawing from regular bronchodilators

Exclusion Criteria:

* Respiratory tract infection (both upper and lower) treated with antibiotics in last 12 weeks
* Clinically significant abnormal values for safety laboratory tests or physical examination
* History or suspected history of drug or alcohol abuse within the past 5 years.
* Known allergy to the study drug or any of the excipients of the formulation.
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) in last 4 weeks or intention to donate blood or blood products during the study.
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than 5 times the drug's half-life, whichever is longer
* Pre-planned surgery or procedures that would interfere with the conduct of the study.
* Employee of the Investigator or study site or family members of the employees or the Investigator.
* History of regular alcohol consumption within last 6 months
* Unable or unwilling to comply fully with the study protocol.
* Mentally or legally incapacitated.
* Unable or unwilling to undergo multiple venepuncture procedures or having poor access to veins suitable for cannulation.
* History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Additional Exclusion Criteria - Healthy Subjects (Parts A and B) only

-Positive test for alcohol or drugs of abuse

Additional Exclusion Criteria - COPD Subjects (Part C) only

* Positive test for alcohol or drugs of abuse prior to randomisation (unless explained by the subject's medication).
* A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
* COPD exacerbation requiring oral steroids within the last 12 months
* A history of one or more hospitalization for COPD in last 12 months
* Evidence of cor pulmonale or clinically significant pulmonary hypertension.
* Other respiratory disorders: Subjects with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnoea, known alpha1-AT deficiency or other active pulmonary diseases.
* Previous lung resection or lung reduction surgery.
* Active participation in a pulmonary rehabilitation program.
* History of chronic uncontrolled disease that the Investigator believes are clinically significant.
* Documented severe cardiovascular disease: angina, recent or suspected myocardial infarction, History of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in last 3 months.
* Major surgery, (requiring general anaesthesia) within last 6 weeks before the screening visit, or will not have fully recovered from surgery, or planned surgery through the end of the study.
* History of significant non compliance in previous investigational studies or with prescribed medications.
* Requires oxygen, even on an occasional basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | From screening until last visit (up to 10 days after last dose)
  Adverse events
Vital signs | Pre-dose, up to 24 hours post last dose and last visit
  Blood pressure and pulse rate
Laboratory safety assessments | Pre-dose, up to 24 hours post last dose and last visit
  Biochemistry, haematology and urinalysis
ECG | Pre-dose, up to 24 hours post last dose and last visit
  ECG
Physical Examination | Pre-dose, 24 hours post last dose and last visit
Holter Monitoring | 24 hours post dose
  Continuous heart monitoring

SECONDARY OUTCOMES:
Pharmacokinetics (trough measurement Blood sampling for RPL554 concentration) | 24 hour profile after first and last dose, trough measurement on Days 2-5 for Parts B and C
  Blood sampling for RPL554 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicines Evaluation Unit, Manchester
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom